CLINICAL TRIAL: NCT00475241
Title: Exposure Therapy for Chronic PTSD: Efficacy and Mechanisms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDA-2-010-06F
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Combat Disorders; Posttraumatic Stress Disorder
Keywords: Combat Disorders; Cortisol; Posttraumatic Stress Disorder (PTSD); Psychophysiology; Therapy; Treatment; Veterans
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Prolonged Exposure and Present Centered Therapy
Who Masked: Outcomes Assessor
Masking Description: Blinded Assessors
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Exposure Therapy (Experimental): Prolonged exposure therapy for PTSD
  Interventions: Behavioral: Prolonged Exposure therapy for PTSD
- Present Centered Therapy (Active Comparator): Present centered therapy for PTSD
  Interventions: Behavioral: Present centered therapy for PTSD

INTERVENTIONS:
Behavioral: Prolonged Exposure therapy for PTSD — exposure-based treatment for PTSD
  Arms: Prolonged Exposure Therapy
Behavioral: Present centered therapy for PTSD — present focused coping and problem solving for PTSD
  Arms: Present Centered Therapy

SUMMARY:
The goals of the proposed research are to produce preliminary evidence of PE with OEF/OIF veterans with PTSD and to examine cognitive, psychophysiological, and neuroendocrine mechanisms of change in PTSD treatment. In brief, 36 OEF/OIF veterans with chronic PTSD or PTSS of at least 3 months duration will be randomly assigned to 15 sessions of either PE or TAU (see below for descriptions of the interventions). All veterans will receive psychobiological assessments at pre treatment, mid treatment, post treatment, 3 months, and 6 months follow-up. Each of these assessments will cover in 2 sessions on separate days and will include interview and self-report of symptoms (i.e., PTSD, depression, and general anxiety severity), self-report of PTSD-related cognitions, psychophysiological (i.e., heart rate, skin conductance, respiration, and end-tidal CO2) assessment during neutral and trauma scripts, and assessment of salivary cortisol during neutral and trauma scripts. Also, on the morning prior to each laboratory assessment, patients will collect salivary cortisol at the moment of waking and 30 and 45 minutes post-walking. In addition to these assessments, patients assigned to PE will collect salivary cortisol during three imaginal exposure sessions (sessions 3, 9, and 15).

DETAILED DESCRIPTION:
Effective treatments for PTSD are available, with exposure therapy (ET) programs, including Prolonged Exposure (PE), having the most empirical evidence for effectiveness (Rothbaum et al., 2000). However, among people receiving treatment for PTSD, many are not receiving psychotherapies with empirically proven efficacy. In one VA VISN, only 10% of PTSD specialist therapists reported using ET routinely (Rosen et al., 2004). They suggested that a lack of training and human resources to provide ET, as well as misconceptions about exposure therapy may drive the deficit. Training efforts would be substantially more cost-effective of the proven treatments could be delivered in group formats. Development and proof of efficacy of a group-based PE would provide far more veterans with access to a treatment that can truly foster recovery from the devastating impact of PTSD. This is a central goal of this proposal.

Little is known about the mechanisms through which PE leads to recovery. Delineation of its mechanisms is a critical step towards the development of treatment refinements to improve effectiveness and efficiency of the treatment. We plan to examine the potential roles of cognitive, psychophysiologic and neuroendocrine factors in symptom improvement. The mechanistic component will provide preliminary data on interactions between cognitive change (increased sense of self-competence and control over negative outcomes), psychophysiological habituation (reduced reactivity to trauma related stimuli), and reduced neuroendocrine sensitivity (reduced hypothalamic-pituitary-adrenal (HPA) axis reactivity). We predict that cognitive change, psychophysiological habituation and reduced HPA reactivity will all be related to symptom improvement with effective treatment.

Thirty-six OEF/OIF veterans with chronic PTSD of at least 3 months duration will be randomly assigned to 15 weeks of twice weekly PE-G or TAU. All veterans will receive psychobiological assessments at pre treatment, mid treatment, post treatment, 3 months and 6 months follow-up. Each of these assessments will include interview and self-report of symptoms (i.e., PTSD, depression, and general anxiety severity), self-report of PTSD-related cognitions, psychophysiological (i.e., heart rate, skin conductance, respiration, and end-tidal CO2) assessment during neutral and trauma scripts, and assessment of salivary cortisol during neutral and trauma scripts. Also, on the morning prior to each laboratory assessment, patients will collect salivary cortisol at the moment of waking and 30 and 45 minutes post-walking. The results from this study will be used as pilot data for VA Merit Award and NIMH R01 applications for larger follow-up studies.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF Veterans with combat related posttraumatic stress disorder (PTSD) or posttraumatic stress symptoms (PTSS) of at least 3 months duration with significant impairment (PSSI greater than or equal to 15).

Exclusion Criteria:

* Any current level of personality disorder or suicidal risk that in the judgment of the investigator makes it unlikely or contraindicated that the patient can adhere to the study regimen.
* Psychosis
* Alcohol or substance dependence in the past 3 months
* Working night-shifts
* Changes to psychoactive medication in the past 8 weeks
* Taking medication that makes HPA axis measures difficult to interpret

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Rauch, PhD, Principal Investigator — VA Ann Arbor Healthcare System
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Sripada RK, Rauch SA, Tuerk PW, Smith E, Defever AM, Mayer RA, Messina M, Venners M. Mild traumatic brain injury and treatment response in prolonged exposure for PTSD. J Trauma Stress. 2013 Jun;26(3):369-75. doi: 10.1002/jts.21813. Epub 2013 May 20. PMID 23696427
- [Derived] Sivakumar RK, Samy W, Pakpirom J, Songthamwat B, Karmakar MK. Ultrasound-guided selective trunk block: Evaluation of ipsilateral sensorimotor block dynamics, hemidiaphragmatic function and efficacy for upper extremity surgery. A single-centre cohort study. Eur J Anaesthesiol. 2022 Oct 1;39(10):801-809. doi: 10.1097/EJA.0000000000001736. Epub 2022 Aug 11. PMID 35950709
- [Derived] Rauch SAM, King AP, Liberzon I, Sripada RK. Changes in Salivary Cortisol During Psychotherapy for Posttraumatic Stress Disorder: A Pilot Study in 30 Veterans. J Clin Psychiatry. 2017 May;78(5):599-603. doi: 10.4088/JCP.15m10596. PMID 28102979

RESULTS

PARTICIPANT FLOW:
Groups:
- Prolonged Exposure: Prolonged exposure therapy for PTSD
  Prolonged Exposure therapy for PTSD: exposure-based treatment for PTSD
Period: Overall Study
Arm/Group | Prolonged Exposure | Present Centered Therapy
Started | 18 | 18
Completed | 11 | 15
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolonged Exposure | Present Centered Therapy | Total
Number analyzed (Participants) | 11 | 15 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (6.5) | 32.9 (7.2) | 31.6 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 9 | 15 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 15 | 26
CAPS [Mean (Standard Deviation); unit: units on a scale] — Clinician Administered PTSD Scale (CAPS) assesses PTSD symptom severity. Scores range from 0 to 136. Higher scores represent more severe symptoms.
  units on a scale | 79.2 (12.1) | 77.4 (12.1) | 78.2 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (Pre & Posttreatment)
Description: Clinician Administered PTSD Scale (CAPS) assesses PTSD symptom severity. Scores range from 0 to 136 and higher scores represent more severe symptoms.
Time Frame: PostTreatment (Week 12)
Population: Treatment Completers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure | Present Centered Therapy
Number analyzed (Participants) | 11 | 15
units on a scale | 30.0 (18.4) | 53.6 (28.7)

2. Secondary Outcome: Trauma Potentiated Startle
Description: Psychophysiological reactivity will be assessed using electromyography collected using a Biopac MP-100 physiology. The potentiation is recorded using a difference score (trauma probe response minus non-trauma probe response).
  The unit of measure is µV. Higher is more response to trauma cue compared to non-trauma cue.
Time Frame: PostTreatment (Week 12)
Population: data was not available due to recording errors for some patients
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Prolonged Exposure Therapy | Present Centered Therapy
Number analyzed (Participants) | 7 | 10
µV | 4.8 (16.2) | 19.5 (30.3)

3. Secondary Outcome: Cortisol Response to Awakening
Description: Area under the curve for awakening, 30 min, and 45 minute salivary cortisol assays.
  Higher means more cortisol response to awakening detected.
Time Frame: PostTreatment (Week 12)
Population: Patient assay quality not adequate for some patients
Measure: Mean (Standard Deviation); unit: min*mg/mL
Arm/Group | Prolonged Exposure | Present Centered Therapy
Number analyzed (Participants) | 7 | 10
min*mg/mL | 1.2 (.4) | .5 (.4)

4. Secondary Outcome: Posttraumatic Cognitions Inventory
Description: Self-report measure of trauma-related cognitions. Range is 21-147. Higher is more problematic trauma-related cognitions.
Time Frame: PostTreatment (Week 12)
Population: patients with missing data not included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure | Present Centered Therapy
Number analyzed (Participants) | 11 | 14
units on a scale | 91.3 (41.9) | 97.1 (45.6)

ADVERSE EVENTS:
Arm/Group | Prolonged Exposure | Present Centered Therapy
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15
Other Adverse Events (participants affected / at risk) | 0/11 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes